CLINICAL TRIAL: NCT01704196
Title: Phase 2, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Trial of Nepicastat for Cocaine Dependence
Brief Title: A Multi-Center Trial of Nepicastat for Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA/VA CS#1031
Record Dates: First submitted 2012-09-17; First posted 2012-10-11 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — nepicastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nepicastat (Active Comparator): Nepicastat 120mg and 100mg riboflavin (once per day) for 11 weeks
  Interventions: Drug: Nepicastat
- Placebo (Placebo Comparator): Placebo capsule containing 100mg riboflavin (once per day) for 11 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nepicastat — 120 mg of active drug and 100mg of riboflavin daily for 11 weeks or matching placebo containing 100mg of riboflavin daily for 11 weeks.
  Arms: Nepicastat
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Nepicastat in improving the number of subjects that achieve abstinence from cocaine and reducing cocaine use in subjects with cocaine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Is seeking treatment for cocaine dependence
* Is able to understand and provide written informed consent
* Has completed all psychological assessments and procedures required during the 7 - 14 day screening period
* If female, agrees to use an acceptable method of birth control
* Is, in the opinion of the Investigator, likely to complete the 11-week Treatment Phase of the study

Exclusion Criteria:

* Please contact the study site for more information

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Matrix Institute on Addictions, Los Angeles, California
  - VA San Diego Healthcare System, San Diego, California
  - VA Medical Center - Denver, CO, Denver, Colorado
  - Mountain Manor Treatment Center at Baltimore, Baltimore, Maryland
  - Pacific Institute for Research and Evaluation, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - Cincinnati Addiction Research Center, Cincinnati, Ohio
  - University of Pennsylvania - Treatment Research Center, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - George E. Wahlen VA Medical Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo capsule containing 100mg riboflavin (once per day) for 11 weeks.
  Placebo
Period: Overall Study
Arm/Group | Nepicastat | Placebo
Started | 90 | 89
Completed | 71 | 65
Not Completed | 19 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepicastat | Placebo | Total
Number analyzed (Participants) | 90 | 89 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (8.2) | 49.0 (8.2) | 49.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 75 | 77 | 152
Region of Enrollment [Number; unit: participants]
  United States | 90 | 89 | 179

OUTCOME MEASURES:

1. Primary Outcome: Abstinence (Weeks 10 - 11)
Description: Number of subjects that abstained from cocaine from weeks 10 through 11
Time Frame: Weeks 10 - 11
Measure: Count of Participants; unit: Participants
Arm/Group | Nepicastat | Placebo
Number analyzed (Participants) | 90 | 89
Participants | 4 | 7

2. Secondary Outcome: Reduction in Use (Weeks 1 - 11)
Description: Proportion of Subjects with a 50% or More Reduction in Cocaine Use from Baseline through week 11
Time Frame: Baseline through week 11
Measure: Number; unit: participants
Arm/Group | Nepicastat | Placebo
Number analyzed (Participants) | 90 | 89
participants | 13 | 20

ADVERSE EVENTS:
Arm/Group | Nepicastat | Placebo
Serious Adverse Events (participants affected / at risk) | 8/90 | 2/89
Other Adverse Events (participants affected / at risk) | 80/90 | 67/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nepicastat (N=90) | Placebo (N=89)
Hospitalization for Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization for Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalization for acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization for Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for depression and suicidality (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for angioedema secondary to lisinopril (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalization for head wounds and cracked ribs (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization for the flu (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization for stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nepicastat (N=90) | Placebo (N=89)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 7 (10)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (5)
Headache (Nervous system disorders) | 16 (20) | 11 (17)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2)
Hypertension (Vascular disorders) | 6 (9) | 7 (9)
Dizziness (Nervous system disorders) | 8 (10) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (5)
Abdominal Discomfort (Gastrointestinal disorders) | 5 (5) | 4 (4)
Toothache (Gastrointestinal disorders) | 7 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 9 (10)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (3)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No